CLINICAL TRIAL: NCT04019743
Title: A Randomized, Open-label, Fasted, Single Dose, Crossover Study to Investigate the Pharmacokinetic Profiles and Safety of CKD-333 in Healthy Volunteers
Brief Title: Clinical Study to Investigate the Pharmacokinetic Profiles and Safety of CKD-333 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A70_07BE1906P
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 1. Period 1: Treatment A
  2. Period 2: Treatment B
  3. Period 3: Treatment C
  Interventions: Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T
- Group 2 (Experimental): 1. Period 1: Treatment C
  2. Period 2: Treatment A
  3. Period 3: Treatment B
  Interventions: Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T
- Group 3 (Experimental): 1. Period 1: Treatment B
  2. Period 2: Treatment C
  3. Period 3: Treatment A
  Interventions: Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T
- Group 4 (Experimental): 1. Period 1: Treatment C
  2. Period 2: Treatment B
  3. Period 3: Treatment A
  Interventions: Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T
- Group 5 (Experimental): 1. Period 1: Treatment B
  2. Period 2: Treatment A
  3. Period 3: Treatment C
  Interventions: Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T
- Group 6 (Experimental): 1. Period 1: Treatment A
  2. Period 2: Treatment C
  3. Period 3: Treatment B
  Interventions: Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T; Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T

INTERVENTIONS:
Drug: CKD-330 16/10mg Tab. 1T and D086 Tab. 1T — single oral administration under fasting condition
  Other Names: Treatment A
Drug: CKD-333 16/10/40mg formulation 1 Tab. 1T — single oral administration under fasting condition
  Other Names: Treatment B
Drug: CKD-333 16/10/40mg formulation 2 Tab. 1T — single oral administration under fasting condition
  Other Names: Treatment C

SUMMARY:
This study is a randomized, open-label, fasted, single dose, crossover study to investigate the pharmacokinetic profiles and safety of CKD-333 in healthy volunteers.

DETAILED DESCRIPTION:
To healthy subjects of twenty-four (24), following treatments are administered dosing in each period and wash-out period is a minimum of 14 days.

Reference drug: 1) CKD-330 16/10mg Tab. 2) D086 Tab. Test drug: 1) CKD-333 16/10/40mg formulation 1 Tab. 2) CKD-333 16/10/40mg formulation 2 Tab.

Pharmacokinetic blood samples are collected up to 72hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 55 years old healthy subject at the screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and a total body weight ≥ 55 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, vital signs, ECG etc.)
5. Individuals who signed an informed consent form approved by the IRB of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational drug
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of study drug infusion
7. Individuals with the ability and willingness to participate during the study period

Exclusion Criteria:

1. Individuals with a medical evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune disease (excluding simple dental history such as dental calculus, impacted tooth, wisdom tooth, etc.)
2. Individuals with a medical history of gastrointestinal disease (e.g., gullet disease including esophageal achalasia, esophagostenosis, or Crohn's disease) or operations (excluding simple appendectomy, herniotomy, or tooth extraction surgery) that may affect drug absorption
3. Individuals with the following laboratory test results:

   * ALT or AST > 2x the upper limit of the normal range
   * CK > 3x the upper limit of the normal range
4. A history of regular alcohol consumption exceeding 210 g/week within the 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Individuals who smoked more than 20 cigarettes per day within 6 months prior to screening
6. Individuals who had been administered investigational product(s) of other clinical study or bioequivalence study within the 6 months prior to the first dose of this study
7. Individuals with the following vital signs results at screening Individuals who had sitting blood pressure ≥90 mmHg or <140 mmHg (systolic) or ≥90 mmHg or <60 mmHg (diastolic)
8. Individuals with a medical history of significant alcohol abuse or drug abuse within one year prior to the screening
9. Individuals who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first dose of investigational product(s)
10. Individuals who had taken prescription or nonprescription drugs within the 10 days prior to the first dose of investigational product(s)
11. Individuals who donated whole blood within the 2 months, or blood components within 1 month prior to the first dose of the investigational product(s)
12. Individuals with severe acute/chronic medical or psychiatric conditions that may increase the risk associated with study participation or investigational product(s) administration, or may interfere with the interpretation of study results
13. Individuals with hypersensitivity to ingredients used in the investigational product(s)
14. Patient with hyperkalemia
15. Patients with hepatopathy
16. Patients with hereditary angioedema, ACE inhibitors or angiotensin Ⅱ receptor antagonists who have a history of angioedema
17. Primary hyperaldosteronism
18. Patients with aortic valve stenosis, mitral (valve) stenosis, hypertrophic obstructive cardiomyopathy
19. Patients with ischemic heart disease, ischemic cardiovascular disease, cerebrovascular disease
20. Patients with Intravascular volume depletion
21. Patients with nephropathy (eGFR<60 ml/min/1.73 m2)
22. Patients with renal artery stenosis
23. Patients with muscle disease
24. Patients with Hypothyroidism
25. Women who are pregnant or may be pregnant
26. Patients with a history of muscle toxicity when using statins or fibrates
27. Patients with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
28. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-28 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-330, D086, CKD-333 | Pre-dose (0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Area under the CKD-330/D086/CKD-333 concentration in blood-time curve from zero to final
Cmax of CKD-330, D086, CKD-333 | Pre-dose (0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  The maximum CKD-330/D086/CKD-333 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: No